CLINICAL TRIAL: NCT02964767
Title: Prevalence of HIV-Tb co Infections Among HIV Patients and Their CD4+ T Cell Status-A Single Centre Study in India
Brief Title: HIV-Tb Confections Among HIV Patients
Status: Completed | Type: Observational
Sponsor: Singh, Ranjan Kumar, M.D. (Individual)
Responsible Party: Principal Investigator, Ranjan Kumar Singh, Nodal officer of ART centre, Sadar Hospital., Singh, Ranjan Kumar, M.D.
Other Study IDs: SinghRK
Record Dates: First submitted 2016-11-05; First posted 2016-11-16 (Estimated); Results first posted 2017-08-07 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-09

CONDITIONS: HIV
Keywords: HIV; HIV-Tb co infection; CD4 Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV mono infection: HIV Patients do not have active Mycobacterium Tuberculosis infection
- HIV-Tb. co infection: Patients with HIV and MycobacteriumTuberculosis co infections

SUMMARY:
A cross sectional study would be done for prevalence of HIV-Tb. co infection among patients of HIV enrolled at ART centre, Khagaria, India, during June' 2015 to May' 2016. A comparative study of CD4 (cluster of differentiation 4) T cell count among HIV-Tb. co infected patient and HIV patients would be taken in account.

DETAILED DESCRIPTION:
Introduction

HIV infection increases the susceptibility of Mycobacterium Tuberculosis (M.Tb.) infection, and hastens its progression due to changes in immune status of the patients. In fact, tuberculosis is now the most common opportunistic infection in patients, who die from AIDS. Immune response in tuberculosis and other infections induces cytokines that enhance replication of HIV, and derives the patient to full blown AIDS. the prevalence of HIV/Tb co-infections have been reported to 0.4% to 20.1% from different regions of northern part of india. India is one of the six countries, those are accounted for 60 percent new cases of tuberculosis, and the BRICS countries collectively account for approximately 50 perce

nt cases of worldwide tuberculosis. The prevalence of multidrug resistant tuberculosis(MDR-TB.) is two-threefold higher in HIV co-infected patients; as HIV infected people rapidly acquire the active disease including resistant strain of M. Tb. and rapidly transmit the disease among population including PLHIV, who in turn, manifest the active drug resistant tuberculosis.

Methods

* This is cohort study among patients of HIV, attending ART (Antiretroviral therapy) center khagaria, Bihar, India during June' 2015 to May' 2016.
* Patients enrolled at the centre were subjected to screening for Mycobacterium tuberculosis infection by doing ESR, mantoux test, chest x-ray, sputum examination for acid fast bacillus (AFB) and nucleic acid amplification test.
* HIV/Tb co infected patients were given cotrimoxazole.
* Patients' data-for example, age, sex, co infection with tuberculosis would be recorded.
* Sputum positivity, radiological features, and extra pulmonary manifestations would be recorded and statistical analysis would be done
* Statistical analysis, such as, mean, standard deviation(SD), student T test, p-values would be done. P-value significance would be measured at p < .05.

ELIGIBILITY:
Inclusion Criteria:

* Patients of HIV+ enrolled ART centre

Exclusion Criteria:

* Lost to follow up patients (LFU)
* Patients died before the treatment started
* Children below 5 years

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV population
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ranjan K Singh, M.D., Principal Investigator — Physician cum nodal officer, ART centre, Khagaria, India.
Locations (1):
- ART centre, Sadar Hospital, Khagaria, Bihar, India

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Festenstein F, Grange JM. Tuberculosis and the acquired immune deficiency syndrome. J Appl Bacteriol. 1991 Jul;71(1):19-30. No abstract available. PMID 1894579
- [Background] Getahun H, Gunneberg C, Granich R, Nunn P. HIV infection-associated tuberculosis: the epidemiology and the response. Clin Infect Dis. 2010 May 15;50 Suppl 3:S201-7. doi: 10.1086/651492. PMID 20397949
- [Background] Global Tuberculosis Report 2016, World Health Organisation, Geneva.
- [Background] Perrin F, Breen R, Lipman M. : HIV and Tuberculosis co-infection. ABC of HIV and AIDS. Michael W, et al (ed): Wiley-Blackwell, BMJ Publishing Group Limited 6:42-47,2012
- Available data/document: Epidemiological report — http://www.who.int
- Available data/document: Clinical Study Report — http://www.Wiley.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with HIV infection enrolled at ART centre, Khagaria, India, during June'2015 to May'2016 were recruited.
Pre-assignment Details: patients, who were Lost to Follow Up (LFU), were excluded from study.
Groups:
- HIV,: HIV mono infected patients,
- HIV/Tb.: Patients with HIV/Tb. co infection
Period: Overall Study
Arm/Group | HIV, | HIV/Tb.
Started | 171 | 48
Completed | 171 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1.HIV: patients with mono HIV infections
- 2.HIV/Tb.: Patients with HIV/Tb. co infections
- Total: Total of all reporting groups
Arm/Group | 1.HIV | 2.HIV/Tb. | Total
Number analyzed (Participants) | 171 | 48 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.26 (12.77) | 34.97 (11.21) | 33.63 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 14 | 94
  Male | 91 | 34 | 125

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of HIV/Tb. co Infections Among Patients of HIV Enrolled at ART Center.
Description: % Prevalence of HIV/Tb. co infections= no.of HIV/Tb. co infection (48)/total no. of enrolled patients of HIV including HIV/Tb. co infections (219) x 100, i.e. 21.9%
Time Frame: 12 months
Measure: Number; unit: participants
Groups:
- Prevalence of HIV/Tb. co Infection: Percentage of Tb. co infections among HIV patients enrolled at ART center.
Arm/Group | Prevalence of HIV/Tb. co Infection
Number analyzed (Participants) | 219
participants | 48

2. Secondary Outcome: Comparing CD4+ T Cell Count in HIV-Tb. and HIV Cases.
Description: CD4 cell counts of HIV patients and HIV/co infection patients would be analysed by student T test, and p value would be estimated.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: cells/µL
Groups:
- 1.HIV: HIV patients only
Arm/Group | 1.HIV | 2.HIV/Tb.
Number analyzed (Participants) | 171 | 48
cells/µL | 314.63 (317.49) | 254.29 (218.19)
Statistical Analysis 1: Comparison: 1.HIV vs 2.HIV/Tb; Test type: Other; p < 0.049, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 months
Description: other opportunistic infections
Groups:
- HIV,: HIV patients
- HIV/Tb. co Infections: Patients with HIV-Tb. co infections
Arm/Group | HIV, | HIV/Tb. co Infections
All-Cause Mortality (participants affected / at risk) | 0/171 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/171 | 0/48
Other Adverse Events (participants affected / at risk) | 6/171 | 2/48
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV, (N=171) | HIV/Tb. co Infections (N=48)
giddiness (Nervous system disorders) | 6 (8) | 2 (6) — caused by ART drug Efavirenz.

LIMITATIONS AND CAVEATS:
this is a cross sectional study; findings are limited to the patients attending ART centre.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No